CLINICAL TRIAL: NCT01190514
Title: Phase 1, Open-Label, Randomized, Single-Dose, 4-Treatment, 4-Period Crossover Bioequivalence Study Comparing 25 Mg and 50 Mg Formulations of DVS-233 SR and Investigate Food Effect on 50 Mg Formulations of DVS-233 SR Tablet Under Fed and Fasted Conditions
Brief Title: Phase 1 Study To Test the Bioequivalence Between Two 25 mg Tablets vs. One 50 mg Tablet Under Fast/Fed Condition and Evaluate Food Effect of Desvenlafaxine Succinate Sustained Release (DVS SR)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B2061035
Record Dates: First submitted 2010-08-24; First posted 2010-08-27 (Estimated); Results first posted 2012-01-27 (Estimated); Last update posted 2012-01-27 (Estimated); Status verified 2011-12

CONDITIONS: Depression - Major Depressive Disorder
Keywords: DVS SR; healthy; Bioequivalence study
MeSH Terms: interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bioequivalence and Food effect (Experimental)
  Interventions: Drug: desvenlafaxine succinate sustained release

INTERVENTIONS:
Drug: desvenlafaxine succinate sustained release — Two tablets of 25 mg, single administration, under fed condition
  Other Names: DVS-233 SR, Pristiq
Drug: desvenlafaxine succinate sustained release — One tablet of 50 mg, single administration, under fed condition
  Other Names: DVS-233 SR, Pristiq
Drug: desvenlafaxine succinate sustained release — Two tablets of 25 mg, single administration, under fast condition
  Other Names: DVS-233 SR, Pristiq
Drug: desvenlafaxine succinate sustained release — One tablet of 50 mg, single administration, under fast condition
  Other Names: DVS-233 SR, Pristiq

SUMMARY:
To determine the bioequivalence of 2 tablets of 25 mg sustained release (SR) formulation of DVS and 1 tablet of 50 mg SR formulation of DVS under fed and fast conditions.

To investigate the effect of high-fat meal on pharmacokinetics of desvenlafaxine after administration of 50 mg SR formulation of DVS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2061035&StudyName=Phase%201%20Study%20To%20Test%20the%20Bioequivalence%20Between%20Two%2025%20mg%20Tablets%20vs.%20One%2050%20mg%20Tablet%20Under%20Fast/Fed%20Condition%20and%20Evaluate%20Food

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants randomized to an open-label treatment sequence beginning in Period 1 with 25 milligrams as 2 tablets (25 mg*2) in fed state=A; or a 50 mg tablet in fed state=B; or 25 mg*2 tablets in fasted state=C; or a 50 mg tablet in fasted state=D in a cross-over, 4-period design. Treatment groups sequenced as: ABCD, BADC, CDAB, and DCBA.
Groups:
- DVS SR 25 mg*2 Fed (A) First: Desvenlafaxine sustained release (DVS SR) formulation (PF-0212375) 25 milligrams (mg) as 2 tablets (25 mg*2) on Day 1 of study period in fed state (finished a high-fat breakfast 20 minutes prior to dosing).
- DVS SR 50 mg Fed (B) First: DVS SR 50 mg tablet on Day 1 of study period in fed state.
- DVS SR 25 mg*2 Fasted (C) First: DVS SR 25 mg*2 tablets on Day 1 of study period in fasted state (fasted 8 hours prior to dosing).
- DVS SR 50 mg Fasted (D) First: DVS SR 50 mg tablet on Day 1 of study period in fasted state.
Period: First Intervention (Period 1)
Arm/Group | DVS SR 25 mg*2 Fed (A) First | DVS SR 50 mg Fed (B) First | DVS SR 25 mg*2 Fasted (C) First | DVS SR 50 mg Fasted (D) First
Started | 11 | 10 | 10 | 10
Completed | 10 (Discontinued participant received treatment A of sequence ABCD.) | 10 | 10 | 10
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Second Intervention (Period 2)
Arm/Group | DVS SR 25 mg*2 Fed (A) First | DVS SR 50 mg Fed (B) First | DVS SR 25 mg*2 Fasted (C) First | DVS SR 50 mg Fasted (D) First
Started | 10 (Period 2 received treatment B) | 10 (Period 2 received treatment A) | 10 (Period 2 received treatment D) | 10 (Period 2 received treatment C)
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention (Period 3)
Arm/Group | DVS SR 25 mg*2 Fed (A) First | DVS SR 50 mg Fed (B) First | DVS SR 25 mg*2 Fasted (C) First | DVS SR 50 mg Fasted (D) First
Started | 10 (Period 3 received treatment C) | 10 (Period 3 received treatment D) | 10 (Period 3 received treatment A) | 10 (Period 3 received treatment B)
Completed | 9 (Discontinued participant received treatments ABC of sequence ABCD.) | 10 | 10 | 10
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Fourth Intervention (Period 4)
Arm/Group | DVS SR 25 mg*2 Fed (A) First | DVS SR 50 mg Fed (B) First | DVS SR 25 mg*2 Fasted (C) First | DVS SR 50 mg Fasted (D) First
Started | 9 (Period 4 received treatment D) | 10 (Period 4 received treatment C) | 10 (Period 4 received treatment B) | 10 (Period 4 received treatment A)
Completed | 9 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Participants randomized to 1 of the 4 treatment sequences beginning with DVS SR 25 mg*2 Fed (A); or DVS SR 50 mg Fed (B); or DVS SR 25 mg*2 Fasted (C); or DVS SR 50 mg Fasted (D).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 37.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to 48 Hours (AUC48)
Description: Area under the plasma concentration versus time curve from time zero (pre-dose) to 48 hours post dose; measured as nanograms multiplied by hours divided by milliliters (ng*hr/mL).
Time Frame: Day 1 of Periods 1, 2, 3, and 4: pre-dose, 0 hour, and 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose
Population: Pharmacokinetic parameter analysis (PK) population: all participants randomized and treated and had at least 1 of the PK parameters of primary interest in at least 1 treatment period. N=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- DVS SR 25 mg*2 Fed: DVS SR 25 mg*2 tablets on Day 1 of study period in fed state.
- DVS SR 50 mg Fed: DVS SR 50 mg tablet on Day 1 of study period in fed state.
- DVS SR 25 mg*2 Fasted: DVS SR 25 mg*2 tablets on Day 1 of study period in fasted state.
- DVS SR 50 mg Fasted: DVS SR 50 mg tablet on Day 1 of study period in fasted state.
Arm/Group | DVS SR 25 mg*2 Fed | DVS SR 50 mg Fed | DVS SR 25 mg*2 Fasted | DVS SR 50 mg Fasted
Number analyzed (Participants) | 41 | 40 | 40 | 39
ng*hr/mL | 2948 (726.28) | 2966 (836.52) | 2632 (764.41) | 2777 (893.35)
Statistical Analysis 1: Comparison: DVS SR 25 mg*2 Fasted vs DVS SR 50 mg Fasted; DVS SR 25 mg*2 fasted (test); DVS SR 50 mg fasted (reference). Natural log transformed AUC48: mixed models analysis with sequence, period, treatment (formulation by food status) as fixed effects and subject within sequence as a random effect; Test type: Non-Inferiority or Equivalence — Bioequivalence of the two treatments was to be concluded if the 90% CIs for the ratio of adjusted geometric means for AUC48 fell wholly within (80%, 125%); Mixed Models Analysis; ratio (%) of adjusted geometric means = 95.56, 90% CI 2-sided [86.94 to 105.04] — Adjusted mean difference and the 90% CI for the difference were exponentiated to provide an estimate of the ratio of adjusted geometric means (test/reference)
Statistical Analysis 2: Comparison: DVS SR 25 mg*2 Fed vs DVS SR 50 mg Fed; DVS SR 25 mg*2 fed (test); DVS SR 50 mg fed (reference). Natural log transformed AUC48: mixed models analysis with sequence, period, treatment (formulation by food status) as fixed effects and subject within sequence as a random effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; ratio (%) of adjusted geometric means = 101.31, 90% CI 2-sided [97.17 to 105.64] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: DVS SR 50 mg Fed vs DVS SR 50 mg Fasted; Food effect DVS SR 50 mg fed (test) versus DVS SR 50 mg fasted (reference). Natural log transformed AUC48: mixed models analysis with sequence, period, treatment (formulation by food status) as fixed effects and subject within sequence as a random effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; ratio (%) of adjusted geometric means = 108.76, 90% CI 2-sided [101.10 to 117.01] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Day 1 of Periods 1, 2, 3, and 4: pre-dose, 0 hour, and 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose
Population: PK population; N=number of participants contributing to the median.
Measure: Median (Full Range); unit: hours
Arm/Group | DVS SR 25 mg*2 Fed | DVS SR 50 mg Fed | DVS SR 25 mg*2 Fasted | DVS SR 50 mg Fasted
Number analyzed (Participants) | 41 | 40 | 40 | 39
hours | 6.00 [4.00 to 12.0] | 8.00 [2.00 to 12.0] | 6.00 [4.00 to 16.0] | 6.00 [4.00 to 24.0]

3. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Cmax measured as nanograms divided by milliliters (ng/mL).
Time Frame: Day 1 of Periods 1, 2, 3, and 4: pre-dose, 0 hour, and 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose
Population: PK population; N=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DVS SR 25 mg*2 Fed | DVS SR 50 mg Fed | DVS SR 25 mg*2 Fasted | DVS SR 50 mg Fasted
Number analyzed (Participants) | 41 | 40 | 40 | 39
ng/mL | 130.6 (29.711) | 131.0 (36.308) | 107.3 (26.773) | 112.1 (28.510)
Statistical Analysis 1: Comparison: DVS SR 25 mg*2 Fasted vs DVS SR 50 mg Fasted; DVS SR 25 mg*2 fasted (test); DVS SR 50 mg fasted (reference). Natural log transformed Cmax: mixed models analysis with sequence, period, treatment (formulation by food status) as fixed effects and subject within sequence as a random effect; Test type: Non-Inferiority or Equivalence — Bioequivalence of the two treatments was to be concluded if the 90% CIs for the ratio of adjusted geometric means for Cmax fell wholly within (80%, 125%); Mixed Models Analysis; Ratio (%) of adjusted geometric means = 95.10, 90% CI 2-sided [89.37 to 101.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DVS SR 25 mg*2 Fed vs DVS SR 50 mg Fed; DVS SR 25 mg*2 fed (test); DVS SR 50 mg fed (reference). Natural log transformed Cmax: mixed models analysis with sequence, period, treatment (formulation by food status) as fixed effects and subject within sequence as a random effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Ratio (%) of adjusted geometric means = 101.30, 90% CI 2-sided [94.66 to 108.40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: DVS SR 50 mg Fed vs DVS SR 50 mg Fasted; Food effect DVS SR 50 mg fed (test) versus DVS SR 50 mg fasted (reference). Natural log transformed Cmax: mixed models analysis with sequence, period, treatment (formulation by food status) as fixed effects and subject within sequence as a random effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; ratio (%) of adjusted geometric means = 115.54, 90% CI 2-sided [108.59 to 122.94] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Terminal Elimination Half-life (t 1/2)
Description: Terminal elimination (plasma decay) half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Day 1 of Periods 1, 2, 3, and 4: pre-dose, 0 hour, and 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose
Population: PK population; N=number of participants contributing to the median.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | DVS SR 25 mg*2 Fed | DVS SR 50 mg Fed | DVS SR 25 mg*2 Fasted | DVS SR 50 mg Fasted
Number analyzed (Participants) | 41 | 40 | 40 | 39
hours | 10.50 (2.2478) | 10.72 (2.8931) | 12.71 (6.0106) | 11.13 (2.9444)

5. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf)
Description: Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: Day 1 of Periods 1, 2, 3, and 4: pre-dose, 0 hour, and 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose
Population: PK population; N=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | DVS SR 25 mg*2 Fed | DVS SR 50 mg Fed | DVS SR 25 mg*2 Fasted | DVS SR 50 mg Fasted
Number analyzed (Participants) | 41 | 40 | 40 | 39
ng*hr/mL | 3171 (820.37) | 3216 (973.36) | 3008 (1147.6) | 3052 (1059.9)

6. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Time of the Last Quantifiable Concentration (AUClast)
Time Frame: Day 1 of Periods 1, 2, 3, and 4: pre-dose, 0 hour, and 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose
Population: PK population; N=number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | DVS SR 25 mg*2 Fed | DVS SR 50 mg Fed | DVS SR 25 mg*2 Fasted | DVS SR 50 mg Fasted
Number analyzed (Participants) | 41 | 40 | 40 | 39
ng*hr/mL | 2948 (726.28) | 2966 (836.47) | 2631 (767.89) | 2778 (894.03)

ADVERSE EVENTS:
Time Frame: Events collected from the time of informed consent up to 28 days after last dose of study treatment.
Description: Same event may appear as both an AE and SAE, however, are presented as distinct events; may be categorized as SAE in 1 subject and as non-SAE in another, or 1 subject may have experienced both an SAE and non-SAE during study. Participants are counted multiple times due to the transition through the cross-over sequences.
Groups:
- DVS SR 25 mg*2 Fed: DVS SR 25 mg*2 tablets on Day 1 of study period in fed state (finished a high-fat breakfast 20 minutes prior to dosing).
- DVS SR 25 mg*2 Fasted: DVS SR 25 mg*2 tablets on Day 1 of study period in fasted state (fasted 8 hours prior to dosing).
Arm/Group | DVS SR 25 mg*2 Fed | DVS SR 50 mg Fed | DVS SR 25 mg*2 Fasted | DVS SR 50 mg Fasted
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40 | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 19/41 | 19/40 | 19/40 | 16/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DVS SR 25 mg*2 Fed (N=41) | DVS SR 50 mg Fed (N=40) | DVS SR 25 mg*2 Fasted (N=40) | DVS SR 50 mg Fasted (N=39)
Eyelid irritation (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 4 | 3 | 3
Hunger (General disorders) | 0 | 0 | 1 | 2
Vessel puncture site haematoma (General disorders) | 1 | 1 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 2 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 4 | 5 | 4
Somnolence (Nervous system disorders) | 5 | 1 | 4 | 2
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Ejaculation delayed (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 1 | 1
Hot flush (Vascular disorders) | 0 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.